CLINICAL TRIAL: NCT02177162
Title: Knee Osteoarthritis Care: A Quality Improvement Intervention in Physiotherapists
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient participants recruited in the intervention group
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: S56904
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2023-01-30 (Actual); Status verified 2016-10

CONDITIONS: Quality of Knee Osteoarthritis Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention= education peer review group (Other): For this controlled trial a group of physiotherapists will recieve specific education about optimal exercise therapy for patioents with knee OA in early stage
  Interventions: Other: Education to physiotherapists

INTERVENTIONS:
Other: Education to physiotherapists

SUMMARY:
Physiotherapists' knee OA care is suboptimal. Exercise therapy including a combination of aerobic, muscle strengthening and functional exercises is not always performed and a lot of treatments are used for which there is no evidence. By a continuing education session and a pop-up in the electronic patient file, this study wants to improve knee OA care by focusing on combined exercise therapy.

The study will be performed in collaboration with Pro-Q-Kine, an independent organization implementing quality improvement in Belgian physiotherapists' care. Besides Pro-Q-Kine the study will be performed in collaboration with two or three software producers of physiotherapists' electronic patient files that reached a national homologation for their respective software packages and covering a large part of the Flemish physiotherapists.

Pro-Q-Kine will organize sessions of continuing education with a focus on optimal knee OA care. These sessions will be performed in LOK-groups (local peer-groups of physiotherapists who meet each other for continuing education). At these sessions the physiotherapists will be asked to take part to the study. A pop-up will be installed in the electronic patient file of the participating physiotherapists, lightening up when physiotherapists register a patient with knee OA. The pop-up includes a short message about optimal knee OA care. The physiotherapists will also receive a script for a query in their electronic patient files in order to extract those patients that initiated a treatment for knee OA between 1 year and 3 months before the therapists received education. These patients will receive a letter of their respective physiotherapists in which they are addressed to take part to the study. An informed consent, patient questionnaire and retour-envelope will be included. There will also be the opportunity to complete the questionnaire electronically with an electronic informed consent. The patient questionnaire will include some background details (such as age and gender) and details about the physiotherapeutic treatments they received for knee OA. The patient questionnaire will be coded with a number, referring to the physiotherapist and to the individual patient (the first patient of the first physiotherapist will be coded as 1.01, the 10th patient of the 14th physiotherapist will be coded as 14.10). Patients' names will not be revealed to the investigators and physiotherapists will not have any access to the completed patients' questionnaires. The general practitioners in the environment of the physiotherapist will (probably) receive a letter from the researchers. This letter will contain information about the importance of referral to a physiotherapist in knee OA care and about knee OA care in general. This letter will also refer to the study that is going on in physiotherapists' care, without details.

Six months after the installation of the pop-up, the physiotherapists will be asked again to perform the query to extract patients out of the electronic patient file that have been treated for knee OA and whose treatment sessions had been started in the period of three months from the installation of the pop-up.

ELIGIBILITY:
Inclusion Criteria:

* patients with knee osteoarthritis, treated by a participating physiotherapist within a predefined period

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Quality of knee osteoarthritis care | 0-6 months